CLINICAL TRIAL: NCT04635826
Title: The Role of Expectancy for Cognitive Enhancement in College Students Using Prescription Stimulants Nonmedically
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Did not receive funding
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Karen Cropsey, Professor of Psychiatry, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: 300006362
Record Dates: First submitted 2020-11-04; First posted 2020-11-19 (Actual); Last update posted 2025-04-07 (Actual); Status verified 2025-04

CONDITIONS: Prescription Stimulants; Expectations; Deception
MeSH Terms: conditions — Deception | interventions — Adderall; Tablets

STUDY DESIGN:
Intervention Model Description: 2 X 2, within-subjects, balanced placebo design
Who Masked: Participant, Investigator
Masking Description: This will be a double-blind study. Research assistants will administer capsules, and based on package labeling, tell the participant if they are being administered Adderall or placebo. However, researchers and participants will be blind to which medication is actually being administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Adderall/Truth (Experimental): Participants will be told they are receiving Adderall and will actually be administered Adderall.
  Interventions: Drug: Adderall 10Mg Tablet
- Adderall/Deception (Experimental): Participants will be told they are receiving Adderall and will actually be administered placebo
  Interventions: Drug: Placebo
- Placebo/Truth (Placebo Comparator): Participants will be told they are receiving placebo and will actually be administered placebo.
  Interventions: Drug: Placebo
- Placebo/Deception (Experimental): Participants will be told they are receiving placebo and will actually be administered Adderall
  Interventions: Drug: Adderall 10Mg Tablet

INTERVENTIONS:
Drug: Adderall 10Mg Tablet — Participants will be administered Adderall
  Other Names: Adderall
  Arms: Adderall/Truth; Placebo/Deception
Drug: Placebo — Participants will be administered placebo
  Arms: Adderall/Deception; Placebo/Truth

SUMMARY:
We propose to evaluate the interaction between expectations of receiving stimulants, neurophysiological activity and enhancement of cognitive performance using fMRI.

DETAILED DESCRIPTION:
Participants will then be randomized in a balanced placebo design (BPD) crossing medication (10 mg of mixed amphetamine salts vs placebo) and expectancy (told active medication vs placebo medication), resulting in 4 different conditions 1) mixed amphetamine salts/told stimulant medication; 2) placebo/told stimulant medication; 3) mixed amphetamine salts/told placebo; and 4) placebo/told placebo). Participants will be assigned to four scanning sessions scheduled one week apart and will experience each condition once counterbalanced across participants. Participants will be administered cognitive tasks in and out of the scanner to determine the effects of medication vs expectancy.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years old
* enrolled as a student at UAB or local college/university
* if female, willing to use adequate birth control or abstain from sexual activity

Exclusion Criteria:

* current or prior head injury
* current or prior psychiatric diagnosis (including ADHD)
* neurological disorder or stroke, hypertension, history of blood or circulation disorders (e.g., anemia or sickle-cell), diabetes, brain or spinal abnormalities
* blood pressure more than 130 systolic and 80 diastolic
* heart rate more than 100 beats per minute
* pregnancy
* current illicit substance use as well as nicotine use
* Alcohol or cannabis use that meets DSM-5 criteria for an alcohol or cannabis use disorder
* Inability to abstain from alcohol or cannabis the night before and day of the scanning session
* Inability to reduce caffeine intake to less than 100 mg on testing days in heavy caffeine users
* claustrophobia
* hearing impairment
* vision impairment that cannot be corrected by MRI-compatible lenses

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
How expectancy will affect cognitive performance | 120 minutes
  Using a balanced placebo design, participants will be either administered mixed amphetamine salts or placebo. Their cognitive performance will be assessed in the MRI scanner. The main outcome measure is how the expectancy of stimulants will affect cognitive performance.
The impact that stimulants vs. placebo have on the neural circuitry | 120 minutes
  Using a balanced placebo design, participants will be either administered mixed amphetamine salts or placebo. Their cognitive performance will be assessed in the MRI scanner. This outcome measure is to determine the impact stimulant administration and expectancy of stimulants have on the neural circuitry that supports sustained attention, inhibitory control, and verbal memory processes.
Determine whether stimulant administration and expectancy for stimulants modify the functional connectivity of brain networks | 120 minutes
  Using a balanced placebo design, participants will be either administered mixed amphetamine salts or placebo. Their cognitive performance will be assessed in the MRI scanner. This outcome measure is to determine whether stimulant administration and expectancy for stimulants modify the functional connectivity of brain networks that support cognitive processes under investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Cropsey, PsyD, Principal Investigator — University of Alabama at Birmingham; David Knight, PhD, Principal Investigator — University of Alabama at Birmingham